CLINICAL TRIAL: NCT05815212
Title: Ranibizumab 0.5 mg for Diabetic Macular Edema With Initial Intensive Treatment in the Real World Clinical Setting in Korea (Rising K)
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CRFB002DKR04
Record Dates: First submitted 2023-04-04; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Diabetic Macular Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Patients with DME

SUMMARY:
This study was a multicenter, non-interventional, retrospective chart review of patients with DME who received ranibizumab 0.5 mg as initial intensive treatment in real-world clinical setting in Korea.

Enrolled patients started receiving ranibizumab between 01 December 2019 and 31 October 2020, with records of receiving at least 3 doses in the first 4 months after starting treatment in the data collected until 30 April 2021. Subsequent dosing interval was determined by the treating physician based on the patient's condition. Data were collected for up to 24 weeks (±2 weeks) from the date of first dose of ranibizumab, including best-corrected visual acuity (BCVA) and optical coherence tomography (OCT) results at Week 24. Subjects were identified by review of patient medical records, and those who met the inclusion/exclusion criteria were enrolled.

The primary objective of this study was to evaluate the effectiveness of ranibizumab in patients with DME who received initial intensive treatment by analyzing the mean change in BCVA using data collected during the 24-week follow-up period. Central subfield thickness (CST), intra-retinal fluid (IRF), sub-retinal fluid (SRF), edema improvement, and Diabetic Retinopathy Severity Scale (DRSS) results were also assessed to further analyze the effectiveness of ranibizumab. The total number of ranibizumab doses administered was obtained to determine the pattern of ranibizumab treatment in real-world clinical setting.

All decisions regarding the clinical management and treatment of patients were made by the treating physician according to real-world routine practice, independently of the study. All data collected in this study were extracted from the patient medical records recorded in the process.

ELIGIBILITY:
Inclusion criteria:

* Aged ≥18 years at the start of ranibizumab treatment
* Diagnosed with diabetes mellitus (type 1 or type 2)
* Diagnosed with diabetic macular edema (DME)
* Vision loss due to DME as judged by treating physician
* Medical records of receiving at least 3 doses in 4 months (initial intensive treatment) since the first dose of ranibizumab between 01 December 2019 and 31 October 2020 (data up to 30 April 2021 were collected)
* Records of BCVA and OCT at baseline and Week 24 (±2 weeks) after treatment with ranibizumab

Exclusion criteria:

* Contraindications to ranibizumab according to local label information
* History of systemic or ocular anti-VEGF therapy or loser photocoagulation in the last 90 days before the first dose of ranibizumab
* History of intraocular or periocular corticosteroids in the last 120 days before the first dose of ranibizumab
* History of vitrectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-04-04 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in BCVA at Week 24 (±2 weeks) | Baseline and Week 24 (±2 weeks)

SECONDARY OUTCOMES:
Mean change from baseline in CST at Week 24 | Baseline and Week 24
Percent change in IRF or SRF status from baseline to Week 24 | Baseline and Week 24
Percentage of patients with ≥5-, ≥10- and ≥15-letter gains from baseline to Week 24 | Baseline and Week 24
Percentage of patients with improved edema from baseline to Week 24 | Baseline and Week 24
Percentage of patients with ≥2-step DRSS improvement from baseline to Week 24 | Baseline and Week 24
Percentage of patients with ≥2-step DRSS worsening from baseline to Week 24 | Baseline and Week 24
Mean change from baseline in BCVA at Week 24 according to the quartile of CST change | Baseline and Week 24
Mean change from baseline in BCVA at Week 24 according to the IRF or SRF status change | Baseline and Week 24
Total number of ranibizumab doses administered during the 24-week follow-up period | 24 weeks
Change from baseline in BCVA at Week 24 for patients with and without prior history of anti-VEGF therapy | Baseline and Week 24
Change from baseline in CST at Week 24 for patients with and without prior history of anti-VEGF therapy | Baseline and Week 24
Percent change in IRF status from baseline to Week 24 for patients with and without prior history of anti-VEGF therapy | Baseline and Week 24
Percent change in SRF status from baseline to Week 24 for patients with and without prior history of anti-VEGF therapy | Baseline and Week 24
Percentage of patients with ≥5-, ≥10- and ≥15-letter gains from baseline to Week 24 for patients with and without prior history of anti-VEGF therapy | Baseline and Week 24
Percentage of patients with ≥15 and ≥30 improvement in CST from baseline to Week 24 for patients with and without prior history of anti-VEGF therapy | Baseline and Week 24
Percentage of patients with ≥2-step DRSS improvement and worsening from baseline to Week 24 for patients with and without prior history of anti-VEGF therapy | Baseline and Week 24
Change from baseline in BCVA at Week 24 according to the quartile of CST change for patients with and without prior history of anti-VEGF therapy | Baseline and Week 24
Change from baseline in BCVA at Week 24 according to the IRF status change for patients with and without prior history of anti-VEGF therapy change | Baseline and Week 24
Change from baseline in BCVA at Week 24 according to the SRF status change for patients with and without prior history of anti-VEGF therapy change | Baseline and Week 24
Total number of ranibizumab doses administered during the 24-week follow-up for patients with and without prior history of anti-VEGF therapy | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Seoul, South Korea